CLINICAL TRIAL: NCT06065514
Title: The Complex Role of the Inflammation Response Following an Acute Myocardial Infarction: the INFINITY (INFlammatIoN amI sTudY)
Brief Title: The Role of Inflammation in Myocardial Infarction
Acronym: INFINITY
Status: Recruiting | Type: Observational
Sponsor: Nicosia General Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other); Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, Andreas Mitsis MD MSc, Principal Investigator, Nicosia General Hospital
Other Study IDs: DD5025
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Infarction
Keywords: STEMI; NSTEMI; Inflammation; Unstable Angina; Cytokines; Adipokines; Prognosis
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Inflammation; Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients Group: The study plans to include 120 consecutive patients above 18 years old presenting with STEMI, NSTEMI, or UA and referred for coronary angiography.
- Control Group: 60 patients will consist of the control group. The patient and control group will be matched at baseline by equating certain clinical characteristics of interest between the exposed and unexposed groups. The control group will consist of individuals to whom the obstructive coronary artery disease would be ruled out either by invasive or non-invasive coronary angiography or by myocardium perfusion SPECT or stress echocardiography.

SUMMARY:
The aim of this research is to study the prognostic role of a selected combination of cytokines and adipokines in patients with myocardial infarction, as well as to determine their role in the development of adverse cardiac remodeling.

DETAILED DESCRIPTION:
After an acute myocardial infarction (AMI) the inflammatory response seems to have a central role and is connected to major adverse outcomes such as ischemia-reperfusion injury, adverse cardiac remodeling, infarct size, and poor prognosis. The concept of monitoring inflammatory markers as predictors of post-myocardial prognosis is gaining more momentum. Finding the appropriate inflammatory biomarker that would serve as a prognostic marker after an AMI and could stratify the risk for adverse outcomes, could be extremely useful.

INFINITY is a multi-center, prospective, observational cohort study, aiming to assess the complex role of inflammation in the post-AMI period. The study plans to include 120 consecutive patients above 18 years old admitted to the four centers participating in the study.

A panel of inflammatory cytokines and adipokines will be recorded. A venous blood sample will be collected on patient admission (H0), 6-12 hours after admission (H6-12), 24-48 hours after admission (H24-48), and at the 30-day visit (D30). Blood will be collected for routine laboratory tests, as well as to measure the levels of the cytokines IL-6, IL-10, IL-18, IL-17, and the adipokines leptin, apelin, and chemerin.

60 carefully selected patients will consist of the control group. The control group will consist of individuals to whom the obstructive coronary artery disease would be ruled out either by invasive or non-invasive coronary angiography or by myocardium perfusion SPECT or stress echocardiography. The patient and control group will be matched at baseline by equating certain clinical characteristics of interest between the exposed and unexposed groups.

The study will test the hypothesis that circulating plasma levels of the above inflammatory biomarkers reflect different clinical manifestations of coronary artery disease and correlate with coronary anatomy, the severity of coronary artery disease, and the prognosis in a 6-month follow-up period. Finally, will investigate whether the integration of the above inflammatory biomarkers into the already established prognostic risk stratification model, GRACE score, could further improve its predictive power.

ELIGIBILITY:
Inclusion Criteria:

1. ACS (ST-ACS, NSTE-ACS, UA) referred for coronary angiography
2. Above 18 years old
3. Consent form obtained

Exclusion Criteria:

1. Chronic Renal Failure (CRF) stage IV (e GFR < 29 ml/min or creatinine > 2 mg/dl)
2. Chronic Liver Disease (CLD) (ALT > 2 times upper normal limit)
3. Chronic Inflammation and/or autoimmune diseases
4. Active Ca
5. Recent CVA (less than 1 month)
6. Recent (within 2 weeks) use of glucocorticoid drugs or immunosuppressive agents
7. Acute or chronic infection, major surgery, or trauma in the last month
8. Previous heart transplantation
9. Poor life expectancy
10. Cardiogenic shock
11. Cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute coronary syndromes (ST-ACS, NSTE-ACS, UA), who underwent coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Mortality | 6-months
  The relationship between the levels of each biomarker (peak H24-48 measurement and area under curve based on the pharmacokinetics of each biomarker based on H0, H6-12, H24-48, and D30 post-enrollment measurements) with all-cause 6-month mortality (cardiac and non-cardiac mortality)

SECONDARY OUTCOMES:
Incidence of heart failure | 6-months
  The relationship between the levels of each biomarker (peak measurement H24-48 and area under curve based on the pharmacokinetics of each biomarker based on measurements H0, H6-12, H24-48, and D30 post-enrollment) with the development of heart failure within a follow-up interval of 6 months after enrollment.
Incidence of MACE | 6-months
  The relationship between the levels of each biomarker (peak measurement H24-48 and area under curve based on the pharmacokinetics of each biomarker based on measurements H0, H6-12, H24-48, and D30 post-enrollment) with 6-month MACEs (non-fatal MI, unplanned repeated revascularization, acute heart failure or angina/ACS requiring rehospitalization, sudden cardiac death).
Change in cytokines and adipokines (pg/mL) | 6-months
  The comparison between the values of the studied biomarkers at the four-time intervals (H0, H6-12, H24-48, D30).
Change in the left ventricular end-diastolic volume index (percent) | 6-months
  Change in the left ventricular end-diastolic volume index (percent) is assessed in patients with myocardial infarction at 6-months follow-up with intermediate assessments at day 7 after onset

OTHER OUTCOMES:
Change in IL-6 | 30-days
  The comparison between the values of IL-6 at the four-time intervals (H0, H6-12, H24-48, D30).
Change in IL-10 | 30-days
  The comparison between the values of IL-10 at the four-time intervals (H0, H6-12, H24-48, D30).
Change in IL-18 | 30-days
  The comparison between the values of IL-18 at the four-time intervals (H0, H6-12, H24-48, D30).
Change in IL-17 | 30-days
  The relationship between the levels of IL-17 (peak H24-48 measurement and area under curve based on the pharmacokinetics of each biomarker based on H0, H6-12, H24-48, and D30 post-enrollment measurements) with all-cause 6-month mortality (cardiac and non-cardiac mortality).
Change in Leptin | 30-days
  The comparison between the values of Leptin at the four-time intervals (H0, H6-12, H24-48, D30).
Change in Apelin | 30-days
  The comparison between the values of Apelin at the four-time intervals (H0, H6-12, H24-48, D30).
Change in Chemerin | 30-days
  The comparison between the values of Chemerin at the four-time intervals (H0, H6-12, H24-48, D30).

CONTACTS AND LOCATIONS:
Overall Officials: George Kassimis, MD, PhD, Principal Investigator — Second Department of Cardiology, Aristotle University of Thessaloniki; Stergios Tzikas, MD, PhD, Study Director — Third Department of Cardiology, Aristotle University of Thessaloniki; Antonios Ziakas, MD, PhD, Study Director — First Department of Cardiology, AHEPA University Hospital, Aristotle University of Thessaloniki; Andreas Mitsis, MD, MSc, Study Director — Nicosia General Hospital
Locations (4):
- Nicosia General Hospital, Nicosia, Cyprus
- Greece (3):
  - 1st University Department of Cardiology - AHEPA University Hospital, Thessaloniki
  - 2nd University Department of Cardiology, Thessaloniki
  - 3rd University Department of Cardiology, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share IPD because the sharing of clinical trial data can increase transparency, improve understanding of individual trials, and facilitate the re-use of the data for secondary research, including meta-analyses of individual participant data (IPD meta-analyses).

REFERENCES:
- [Background] Mitsis A, Kadoglou NPE, Lambadiari V, Alexiou S, Theodoropoulos KC, Avraamides P, Kassimis G. Prognostic role of inflammatory cytokines and novel adipokines in acute myocardial infarction: An updated and comprehensive review. Cytokine. 2022 May;153:155848. doi: 10.1016/j.cyto.2022.155848. Epub 2022 Mar 14. PMID 35301174